CLINICAL TRIAL: NCT00730483
Title: Treatment of Patients With Hepatic Neuroendocrine Metastases Using Drug-Eluting Bead Embolization
Brief Title: Doxorubicin Beads in Treating Patients With Unresectable Liver Metastases From Neuroendocrine Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High incidence of biloma and liver abscess after TACE
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeff Geschwind, Professor of Radiology and Oncology, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0739 CDR0000601054; JHOC-J7039; JHOC-NA_000010736; JHOC-SKCCC-J7039
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Tumor; Metastatic Cancer
Keywords: liver metastases; metastatic gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; islet cell carcinoma; gastrinoma; insulinoma; glucagonoma; pancreatic polypeptide tumor; somatostatinoma
MeSH Terms: conditions — Adenoma, Islet Cell; Neoplasm Metastasis; Carcinoma, Islet Cell; Gastrinoma; Insulinoma; Glucagonoma; Somatostatinoma | interventions — Doxorubicin

ARMS (1):
- DEB-TACE (Experimental): PVA microporous hydrospheres loaded with doxorubicin hydrochloride used for the treatment of unresectable liver metastases from neuroendocrine tumors.
  Interventions: Drug: PVA microporous hydrospheres/doxorubicin hydrochloride

INTERVENTIONS:
Drug: PVA microporous hydrospheres/doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Infusing doxorubicin beads into the liver, and blocking blood flow to the tumor, may keep doxorubicin near the tumor and kill more tumor cells.

PURPOSE: This clinical trial is studying the side effects of doxorubicin beads and to see how well they work in treating patients with unresectable liver metastases from neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To gather preliminary data and determine the feasibility of a randomized study of patients with unresectable hepatic neuroendocrine metastases using PVA microporous hydrospheres/doxorubicin hydrochloride.

OUTLINE: A catheter is placed into the right or left hepatic artery. Patients with unifocal tumors will have the catheter or microcatheter placed more selectively into the 2nd or 3rd order branch off the right or left hepatic artery in closer proximity to the tumor. Polyvinyl alcohol (PVA) microporous hydrospheres/doxorubicin hydrochloride mixture is injected into the delivery area.

Patients with less than 75% necrosis at 1 month undergo a second (and possibly a third a month later) chemoembolization.

After completion of study therapy, patients are followed at 1 month, every 2 months for 1 year, and then every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of hepatic neuroendocrine metastases not suitable for radical therapies (e.g., resection or liver transplantation)

  * Histologically proven neuroendocrine tumor
  * Tumors are hypervascular based on visual estimation by investigator
* Predominant to the liver disease, but extrahepatic disease is not an exclusion

  * No predominant extrahepatic liver disease
  * No significant life-threatening extrahepatic disease, in the judgment of the physician
* Recent-interval progression of hepatic liver metastases
* No diffuse hepatic neuroendocrine metastases defined as massive ill-defined tumor involvement measuring > 90% tumor burden

Exclusion criteria:

* Clinically evident ascites (a radiographic finding of trace ascites on imaging is acceptable)
* Complete occlusion of the entire portal venous system
* Evidence of cirrhosis or portal hypertension
* Vascular resistance peripheral to the feeding arteries precluding passage of PVA microporous hydrospheres/doxorubicin hydrochloride

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Must have preserved liver function (Child-Pugh class A-B) without significant liver decompensation

  * No advanced liver disease (e.g., Child-Pugh C class or active gastrointestinal bleeding, encephalopathy, or ascites [trace ascites is acceptable]), meeting the following criteria:

    * Bilirubin > 3 mg/dL
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase > 5 times upper limit of normal
    * Serum creatinine > 2.0 mg/dL
    * Albumin ≤ 2.0 g/dL
* No vascular anatomy or blood that precludes catheter placement or emboli injection
* No presence of arteries supplying the lesion not large enough to accept PVA microporous hydrospheres/doxorubicin hydrochloride
* No collateral vessel pathways potentially endangering normal territories during embolization
* No feeding arteries smaller than distal branches from which they emerge
* Not pregnant

Exclusion criteria:

* See Disease Characteristics
* Another active primary tumor
* Any contraindication for hepatic embolization procedures, including any of the following:

  * Porto-systemic shunt
  * Hepatofugal blood flow
  * Impaired clotting tests (i.e., platelet count < 50,000/mm³, international normalized ratio (INR) ≥ 1.8, or partial thromboplastin time (PTT) ≥ 39 seconds)
  * Renal failure
  * Severe peripheral vascular disease precluding catheterization
* Any contraindication for doxorubicin hydrochloride administration (i.e., serum bilirubin > 5 mg/dL or leukocyte count < 1,500 cells/mm³)
* Allergy to contrast media
* Intolerant to occlusion procedures
* Presence of end arteries leading directly to cranial nerves
* Presence or likely onset of hemorrhage
* Presence of severe atheromatous disease

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Prior anticancer therapy for hepatic neuroendocrine metastases, except previous surgical therapy
* Any continuing complication or prior cancer therapy that has not improved or resolved prior to 21 days before start of treatment, if the investigator determines that the continuing complication will compromise the safety of the patient after treatment with PVA microporous hydrospheres/doxorubicin hydrochloride
* Presence of patent extra-to-intracranial anastomoses or shunts
* Use of PVA microporous hydrospheres/doxorubicin hydrochloride in the following applications:

  * Embolization of large-diameter arteriovenous shunts
  * Pulmonary arterial vasculature
  * Any vasculature where the use of PVA microporous hydrospheres/doxorubicin hydrochloride could pass directly into the internal carotid artery or the above-listed vessels
* Concurrent enrollment in another clinical study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F. Geschwind, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Bhagat N, Reyes DK, Lin M, Kamel I, Pawlik TM, Frangakis C, Geschwind JF. Phase II study of chemoembolization with drug-eluting beads in patients with hepatic neuroendocrine metastases: high incidence of biliary injury. Cardiovasc Intervent Radiol. 2013 Apr;36(2):449-59. doi: 10.1007/s00270-012-0424-y. Epub 2012 Jun 22. PMID 22722717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 patients were enrolled on this protocol at Johns Hopkins University. This study was terminated early due to high incidence of bilomas in patients receiving TACE treatment.
Groups:
- Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE): Patients were treated with DEB-TACE loaded with doxorubicin up to four procedures in 6 months as indicated, for a maximum of six procedures during the course of 2 years. Follow-up clinical examinations, laboratory assessments, and imaging took place 1 month after each DEB-TACE treatment and then every 2 to 3 months for a period of 2 years. Each DEB-TACE procedure used a maximum of 100mg doxorubicin loaded onto 100-300um LC Beads.
Period: Overall Study
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Started | 13
1 Month After First DEB-TACE | 13
6 Months After First DEB-TACE | 10
Completed (12 months after first DEB-TACE) | 6
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 64 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of CTCAE v3.0 Events 1 Month Post DEB-TACE
Description: Safety was assessed at each DEB-TACE procedure and at every follow-up thereafter according to National Cancer Institute Common Toxicity Criteria (CTCAE) v3.0. The study was prematurely terminated due to high incidence of biloma and liver abscess. Safety data below is based off of 13 patients enrolled on protocol at 1 month post initial treatment.
Time Frame: 1 month after initial DEB-TACE treatment
Measure: Number; unit: number of adverse events
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 13
number of adverse events
  Anemia | 1
  Lymphopenia | 2
  Hypotension | 1
  Edema | 2
  Increased INR | 2
  Fatigue | 9
  Fever | 4
  Night sweats | 6
  Alopecia | 3
  Dry skin | 1
  Ascites | 1
  Anorexia | 5
  Biloma | 6
  Constipation | 1
  Diarrhea | 1
  Nausea | 1
  Taste alteration | 1
  Hematoma | 1
  Increased ALT | 5
  Increased AST | 5
  Increased AP | 8
  Hyperbilirubinemia | 1
  Hypoalbuminemia | 5
  Liver abscess | 1
  Hyperglycemia | 5
  Hyponatremia | 1
  Neuropathy | 1
  Abdominal nonspecific pain | 5
  Right upper quadrant pain | 6
  Pain - other | 1
  Dyspnea | 1
  Dyspnea on exertion | 1

2. Secondary Outcome: Tumor Response (Efficacy) - by Response Evaluation Criteria in Solid Tumors (RECIST) and the European Association for the Study of the Liver (EASL) Criteria
Description: Study was terminated and full outcome not assessed. The results below are based on 13 patients at 1 month post DEB-TACE, 10 patients at 6 months, and 6 patients at 12 months.
  RECIST:
  Complete Response (CR): Disappearance of all targeted lesions Partial Response (PR): At least 30% decrease in the sum of longest diameter (LD) of targeted lesions Progressive Disease (PD): At least 20% increase in the sum of LD of targeted lesions Stable Disease (SD): Cases that are not applicable for PD or PR.
  EASL:
  CR: Absence of any enhancement in target lesion PR: Greater than 50% decrease from baseline enhancement in target lesion PD: Greater than 25% increase in target lesion SD: All other cases
Time Frame: 12 months
Population: 13 patients were analyzed for 1 month post-treatment; 10 patients for 6 months post-treatment; and 6 patients at the 12 month post-treatment time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 13
Participants
  RECIST 1 month post-TACE: Complete Response (CR) | 0
  RECIST 1 month post-TACE: Partial Response (PR) | 0
  RECIST 1 month post-TACE: Stable Disease (SD) | 13
  RECIST 1 month post-TACE: Progressive Disease | 0
  EASL 1 month post-TACE: Complete Response (CR) | 0
  EASL 1 month post-TACE: Partial Response (PR) | 8
  EASL 1 month post-TACE: Stable Disease (SD) | 5
  EASL 1 month post-TACE: Progressive Disease | 0
  RECIST 6 months post-TACE: number analyzed (Participants) | 10
  RECIST 6 months post-TACE: Complete Response (CR) | 0
  RECIST 6 months post-TACE: Partial Response (PR) | 1
  RECIST 6 months post-TACE: Stable Disease (SD) | 8
  RECIST 6 months post-TACE: Progressive Disease | 1
  EASL 6 months post-TACE: number analyzed (Participants) | 10
  EASL 6 months post-TACE: Complete Response (CR) | 1
  EASL 6 months post-TACE: Partial Response (PR) | 3
  EASL 6 months post-TACE: Stable Disease (SD) | 6
  EASL 6 months post-TACE: Progressive Disease | 0
  RECIST 12 months post-TACE: number analyzed (Participants) | 6
  RECIST 12 months post-TACE: Complete Response (CR) | 0
  RECIST 12 months post-TACE: Partial Response (PR) | 1
  RECIST 12 months post-TACE: Stable Disease (SD) | 4
  RECIST 12 months post-TACE: Progressive Disease | 1
  EASL 12 months post-TACE: number analyzed (Participants) | 6
  EASL 12 months post-TACE: Complete Response (CR) | 2
  EASL 12 months post-TACE: Partial Response (PR) | 1
  EASL 12 months post-TACE: Stable Disease (SD) | 3
  EASL 12 months post-TACE: Progressive Disease | 0

3. Secondary Outcome: Survival
Description: Survival outcomes not assessed due to premature termination of study.
Time Frame: overall survival
Groups:
- Single Arm: PVA microporous hydrospheres/doxorubicin hydrochloride
Arm/Group | Single Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Biochemical Response - Time to Progression
Description: Biochemical response not assessed due to premature termination of study.
Time Frame: Time to progression, 12 months
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 0

5. Secondary Outcome: Symptomatic Response by Assessing Symptom Severity in Patients
Description: Symptomatic response not assessed due to premature termination of study.
  Scoring system for assessing symptom severity in patients with neuroendocrine/carcinoid syndrome was as follows:
  1. - No symptoms - Patient completely asymptomatic
  2. - Mild symptoms - Patient with symptoms of diarrhea, flushing, or asthma up to 4 times weekly
  3. - Symptoms impact daily living - symptoms of diarrhea, flushing, or asthma up 5-7 weekly
  4. - Severe symptoms - multiple daily symptoms of diarrhea, flushing, or asthma; symptoms require significant reorganization of daily activities
  5. - Disabling symptoms - Patient disabled by multiple attacks and severe symptoms; unable to leave home or requires hospitalization
Time Frame: Duration of study participation, average of 12 months
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 7/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE) (N=13)
Liver biloma requiring drainage (Gastrointestinal disorders) | 4 (4)
Gastric varices (Gastrointestinal disorders) | 1 (1)
Liver abscess (Hepatobiliary disorders) | 2 (2)
Biliary stricture (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE) (N=13)
Abdominal pain (Gastrointestinal disorders) | 9 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 6 (8)
Anxiety (Psychiatric disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pain - coccyx (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased vision (Eye disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema - bilateral extremities (General disorders) | 3 (3)
Elevated ALT (Investigations) | 10 (14)
Elevated alkaline phosphatase (General disorders) | 11 (20)
Elevated AST (Investigations) | 11 (15)
Elevated INR (Investigations) | 5 (5)
Fatigue (General disorders) | 13 (27)
Fever (General disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Pain - general (General disorders) | 2 (2)
Edema - hands (General disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 2 (4)
Hyperglycemia (Investigations) | 9 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left eye swelling (Eye disorders) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytopenia (Blood and lymphatic system disorders) | 1 (2)
Lymphopenia (Investigations) | 4 (5)
Nausea (Gastrointestinal disorders) | 5 (8)
Neuropathy (Nervous system disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (12)
Palpitations (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Right flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes